CLINICAL TRIAL: NCT01252290
Title: Modulation of Breast Cancer Risk Biomarkers in Postmenopausal Women by High Dose Omega-3 Fatty Acids
Brief Title: Breast Cancer Risk Biomarkers in Postmenopausal Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Carol Fabian, MD (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor-Investigator, Carol Fabian, MD, Professor, Director Breast Cancer Prevention Unit, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 12350
Record Dates: First submitted 2010-11-23; First posted 2010-12-02 (Estimated); Results first posted 2016-12-16 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Omacor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lovaza™ (Experimental): Lovaza™ (two 1 gram capsules twice daily) for six months
  Interventions: Drug: Lovaza™

INTERVENTIONS:
Drug: Lovaza™ — 4 capsules daily for 6 months
  Other Names: esters of EPA and DHA

SUMMARY:
This study is designed to gather information on how the prescription drug Lovaza™ which contains omega-3 fatty acids, affects blood and tissue risk biomarkers for breast cancer. This drug is currently approved by the FDA for reducing blood levels of triglycerides.

DETAILED DESCRIPTION:
The central hypothesis is that 6 months of administration of high dose omega-3 fatty acid esters [eicosapentaenoic acid (EPA) 1860 mg, and docosahexaenoic acid (DHA) 1500 mg] daily in the form of a standard prescription strength dose of Lovaza™ (two 1 gram capsules twice daily) will have a favorable side effect profile and potential efficacy as demonstrated by favorable modulation of one or more blood and breast tissue risk biomarkers for breast cancer in postmenopausal women.

ELIGIBILITY:
Inclusion Criteria

* Subjects must be postmenopausal and between the ages of 25 and 69 years. Menopause is defined by no menstrual period for more than one year and intact uterus and ovaries, or women with intact ovaries but without a uterus and age 50 and over, or a woman with both estradiol and follicle stimulating hormone (FSH) in the postmenopausal range or any woman who has had her ovaries removed.
* Subjects must be at increased risk for breast cancer on the basis of at least one of the following criteria:

  * A five-year Gail risk of ≥ 1.67% or ≥ 2X the average risk for a woman of the same age using either the Surveillance Epidemiology and End Results (SEER, http://seer.cancer.gov) database, the NCI Breast Cancer Risk Assessment Tool (www.cancer.gov/bcrisktool), or the International Breast Cancer Intervention Study (IBIS) Risk Evaluator (http://www.emstrials.

org/riskevaluator/), or a ten-year Tyrer-Cuzick model risk of 2x that of the population risk.

* A first degree relative with breast cancer under the age of 60 or multiple second degree relatives with breast cancer.
* Multiple prior biopsies or at least one prior biopsy exhibiting atypical hyperplasia (AH), lobular carcinoma in situ (LCIS), ductal carcinoma in situ (DCIS).
* Random periareolar fine needle aspiration (RPFNA) evidence of hyperplasia with atypia within the last three years;
* Chest or neck radiation before age 30;
* Mammographic breast density by visual estimate equals or exceeds 50%.

  * Subjects must be willing to continue the same hormonal milieu present at baseline throughout trial (Cannot start or stop any type of hormone replacement therapy with the exception of vagifem or estring).
  * Six months or more must have elapsed from completion of a prevention intervention trial (with exception of a weight reduction trial), ingestion of a selective estrogen receptor modulator (SERM) or aromatase inhibitor (AI) prior to baseline biomarker assessment. .
  * Subjects with a history of AH, LCIS, or ER-positive DCIS by diagnostic biopsy, must have been counseled about appropriate standard prevention therapies such as tamoxifen or raloxifene and are either not eligible or are not interested in standard prevention therapies. Women with DCIS must have had appropriate local therapy (lumpectomy plus radiation or mastectomy). If subject has had a DCIS, at least two months must have elapsed from surgery and/or radiation therapy to the involved breast. Only the contra-lateral (uninvolved breast) will be studied by RPFNA. The subject may not have had any radiation therapy to the contra-lateral breast to be studied
  * Subjects must have had a screening mammogram within 6 months of entering the interventional portion of the study and read as not suspicious for breast cancer or if suspicious must have completed all suggested tests including biopsy and found to have no evidence of cancer. Women must be willing to have an off-study mammogram performed 6 months after study entry.
  * Subjects must have had an RPFNA of the breast within six months prior to entering the intervention portion of the study and be willing to have another RPFNA at ~6.5 months after starting Lovaza™.
  * Tissue Eligibility: Subjects must have cytomorphologic evidence of hyperplasia with atypia or borderline atypia (Masood score > 13). There must be ≥500 epithelial cells on the slide for cytomorphology. There must be sufficient reserved methanol-formalin- fixed material for quantitative reverse transcription polymerase chain reaction (RT-qPCR). Frozen tissue must also have been obtained for fatty acid analysis, reverse phase proteomics, adipokines and cytokines, and RT-qPCR.
  * Subjects must be willing to undergo phlebotomy at baseline and 6 months and 6.5 months. Approximately 3 tablespoons of blood will be obtained at baseline and 6 months and 6.5 months or 6 tablespoons if the subject decides to participate in the optional monocyte cytokine release assay .
  * Subjects must produce a spot urine sample at baseline, 6 months, and at study conclusion
  * Subjects must be willing to undergo measurement of height, weight, and BMI and undergo body composite analysis (DEXA) at initiation and conclusion of intervention.
  * Subjects must be willing to complete questionnaires regarding diet and supplement use, quality of life as well as relevant family history personal health and reproductive history and medications at initiation and conclusion of the intervention. Subjects must be willing to sign an informed consent for the entire study and separate consent for repeat RPFNA.

Exclusion Criteria

* Women that have had a metastatic malignancy of any kind.
* Women that have had prior invasive breast cancer, diagnosed or treated within the past five years.
* Women who are currently taking anticoagulants.
* Women who have breast implants.
* Women who have undergone change in their hormonal milieu in the past 6 months.
* Women who have taken omega 3 fatty acid or flaxseed supplements within 3 weeks prior to their baseline RPFNA or women who have taken high dose omega 3 within the past three months.
* Women who regularly take NSAIDS (>7 tablets weekly).
* Women who have taken a SERM, aromatase inhibitor or participated in a chemoprevention or other investigational drug study within six months prior to baseline RPFNA.
* Women who have abnormal renal or hepatic function at baseline, defined as blood chemistry values clinically significantly outside of normal institutional ranges.
* Women who have a history of an allergy, including hives, to fish products.
* Women who have a BMI of 40 kg/m^2 or greater.

Inclusion of Women and Minorities This study utilizes women at increased risk for breast cancer. Subjects recruited from an established cohort of women followed in the Breast Cancer Prevention Center. From previous trials we can expect 6% minority accrual which is similar to our hospital demographics. Males are not included due to the low absolute risk of breast cancer, and the difficulty of performing RPFNA on the male breast.

Ages: 25 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2010-11; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol Fabian, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No
Summary results for the cohort have been published.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lovaza™
Started | 35
Completed | 34
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Lovaza™
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.2 (8.4)
Gender [Count of Participants; unit: Participants]
  Female | 35
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 35
Weight [Mean (Standard Deviation); unit: kilograms] | 71 (14)
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 26.2 (4.7)
5-Year Gail Risk [Mean (Standard Deviation); unit: percent probablity of breast cancer] — Gail Model is one of the models developed to quantify a woman's risk of developing breast cancer. The model incorporates a series of questions related to breast cancer risk factors. Women who have a percentage of risk of 1.66 or higher have a higher than average risk for developing breast cancer.
  Measure taken on 27 participants. Eight participants risk could not be calculated because the model does not allow calculation for women with prior ductal carcinoma in situ (DCIS), lobular carcinoma in situ (LCIS), or invasive breast cancer.
  percent probablity of breast cancer | 3.4 (1.5)

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Subjects That Complete Intervention of Lovaza™ 4 Grams Per Day
Description: To determine the feasibility of an intervention of Lovaza™ 4 grams per day (~ 1800 mg EPA and 1500 mg DHA) administered for 6 months to post-menopausal women under the age of 50.
Time Frame: 6 month visit
Measure: Number; unit: proportion of enrolled participants
Arm/Group | Lovaza™
Number analyzed (Participants) | 34
proportion of enrolled participants | 0.97

2. Secondary Outcome: Modulation of the Risk Biomarker Masood Score
Description: Change in the semiquantitative cytology index score (Masood score) from baseline to end of study. Masood Score range 6 - 24; increasing values denote increasing cytologic abnormality. Thus, negative values for change reflect an improvement, i.e., less cytologic abnormality after intervention.
Time Frame: 6 month value compared to baseline value
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Lovaza™
Number analyzed (Participants) | 34
units on a scale | -1 [-2 to 1]

3. Secondary Outcome: Change in (DHA+EPA):AA Ratio for Phospholipids in Plasma
Description: Change (from baseline to end of study) for the ratio derived from levels of DHA, EPA, and AA (measured as percent of total fatty acid content) in the phospholipid compartment of plasma.
Time Frame: Change from Baseline to Month 6
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Lovaza™
Number analyzed (Participants) | 34
ratio | 0.62 [0.43 to 1.04]

4. Secondary Outcome: Change in Quality of Life
Description: Change in score on Breast Cancer Prevention Trial (BCPT) Symptom Checklist. Summation score of degree of difficulty (scored 0 to 4 each) with 43 individual activities. Thus total score ranges from 0 to 172. Increasing score represents increasing problems with side effects.
Time Frame: Change from Baseline to Month 6
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Lovaza™
Number analyzed (Participants) | 34
units on a scale | 10 [1 to 57]

5. Secondary Outcome: Change in Ki-67 Expression
Description: Immunocytochemical staining for Ki-67 antibody. Percent of 500 benign breast epithelial cells scored that are classified as positively staining.
Time Frame: 6 month value compared to baseline value
Measure: Median (Inter-Quartile Range); unit: change in percent Ki-67 expression
Arm/Group | Lovaza™
Number analyzed (Participants) | 34
change in percent Ki-67 expression | -0.4 [-2.1 to 0]

ADVERSE EVENTS:
Time Frame: duration of intervention, planned at 6 months
Arm/Group | Lovaza™
Serious Adverse Events (participants affected / at risk) | 2/35
Other Adverse Events (participants affected / at risk) | 14/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lovaza™ (N=35)
Ductal carcinoma in situ (Reproductive system and breast disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lovaza™ (N=35)
acid reflux (Gastrointestinal disorders) | 3 (3) — gastric reflux, including gastroesophageal reflux disease
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Breast biopsy (Reproductive system and breast disorders) | 2 (5) — One each LCIS and intraductal papilloma
Diarrhea (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Urinary tract infection (Renal and urinary disorders) | 2 (2)
Breast pain (Reproductive system and breast disorders) | 2 (2)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes